CLINICAL TRIAL: NCT01866566
Title: Phase 4 Study of Live Attenuated Varicella Vaccine After the 2 Doses Vaccination
Brief Title: The Safety and Immunogenicity Research of Live Attenuated Varicella Vaccine After the 2 Doses Vaccination
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BJCDPC-9
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-05

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HBV-3 (Placebo Comparator): one dose HBV
  Interventions: Biological: HBV-3
- HBV-6 (Placebo Comparator): one dose HBV
  Interventions: Biological: HBV-6
- varicella-3 (Experimental): 2 doses varicella vaccine either BCHT or Kengen and 3 month of the interval time
  Interventions: Biological: varicella-3
- varicella-6 (Experimental): 2 doses varicella vaccine either BCHT or Kengen and 6 month of the interval time
  Interventions: Biological: varicella-6

INTERVENTIONS:
Biological: HBV-3 — Give a single 0.5 mL HBV and get blood samples at 0,1.5,4.5 month
  Arms: HBV-3
Biological: HBV-6 — Give a single 0.5 mL HBV and get blood samples at 0,1.5,7.5 month
  Arms: HBV-6
Biological: varicella-3 — Give 2 doses varicella vaccine (a single 0.5 mL) and get blood samples at 0,1.5,4.5 month
  Arms: varicella-3
Biological: varicella-6 — Give 2 doses varicella vaccine (a single 0.5 mL) and get blood samples at 0,1.5,7.5 month
  Arms: varicella-6

SUMMARY:
Through evaluating the immunogenicity and safety for Varicella vaccine two doses immune procedure we could supply scientific and practical evidence for this two doses immune procedure promotion and management.

DETAILED DESCRIPTION:
Healthy participants aged 1 to 12 years old who had never received Varicella Vaccine are divided into three age groups, 1 to 3 years old group, 4 to 6 years old group and 7-12 years old group. In each age group, participants are randomly divided into experiment group and control groups.

ELIGIBILITY:
Inclusion Criteria:

-Participants from Shanxi province are between 1-12 years old are in good healthy determined through medical inquiry, physical examination, clinical judgment of the investor.

Exclusion Criteria:

1. Having a fever (axillary temperature>37.0℃) before enrollment;
2. Having a disease history of seizures, brain disease and the vaccination history of allergies and convulsions;
3. Antibiotics allergy;
4. Having a problem of intramuscular injection because thrombocytopenia or other blood coagulation disorder;
5. Having immunodeficiency or under immunosuppression therapy, radiation therapy;
6. Having respiratory diseases, acute infection, chronic disease and HIV infection;
7. Having systemic skin rash, skin tinea, herpes;
8. Chronic liver and kidney disease;
9. Heart disease, and severe hypertension;
10. Have received whole blood, plasma or immunoglobulin therapy 3 months before enrollment;
11. Have received other live attenuated vaccine vaccination in 30 days before enrollment;
12. Had been infected with Varicella virus and displayed symptom;
13. Have received one or two dose of Varicella vaccine before enrollment;
14. Congenital malformations, growth disorders such as Down's syndrome, diabetes, sickle cell anemia and nervous disorders
15. Guillain-barre syndrome
16. Thyroid resection history or thyroid disease treatment in the past 12 months;
17. Asthma
18. Have participated in other clinical research;
19. Have serious adverse reactions after vaccination, such as allergies, hives, breathing difficulties, angioneurotic edema.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1800 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Antibody titer after 2 doses lived attenuated varicella vaccination | 1 year
  Serums are collected from all participants before and 42 days after the first vaccination, and also 42 days after the second vaccination. The antibody titer to Varicella was detected through FAMA test.

SECONDARY OUTCOMES:
Number of participants who have adverse reaction | 1 year
  The safety is evaluated by systemic and local reaction after each vaccination.

OTHER OUTCOMES:
Number of participants who catch chickenpox | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Nianmin Shi, Study Chair — Beijing Chaoyang District Centers for Disease Control and Prevention
Locations (1):
- Shanxi Centers for Disease Control and Prevention, Yuncheng, Shanxi, China